CLINICAL TRIAL: NCT06503705
Title: Qualitative Investigation Into the Obstacles and Facilitators to the Treatment of Police Officers With Mental Health Disorders
Brief Title: Obstacles and Facilitators to the Treatment of Police Officers With Mental Health Disorders
Acronym: BASP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9140
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorders
Keywords: Mental Disorders; Behavior Disorders; Anxiety Syndrome; Depression Syndrome; Mental health difficulties; Policmen
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Police officers are subject to various professional risk factors that can contribute to the occurrence of mental health difficulties such as depression, anxiety, and post-traumatic stress disorder. In previous work, low use of specialized care structures was noted. Added to this is the carrying of a weapon which represents an element facilitating the passage to self-aggressive action.

The objective of the study is to identify and describe the barriers and facilitators to the treatment of police officers facing mental health difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Be an active, administrative police officer, or scientific and technical police officer of the national police in France for more than a year,
* Or work for the Ministry of the Interior as support staff, or medical staff,
* Agree to participate in the study,
* Agree to talk about the problem without managerial or union preconceptions.

Exclusion Criteria:

* Be in post for the Ministry of the Interior for less than a year.
* Be stationed in the Bas Rhin department (France), where the principal investigator works.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active major subjet, administrative police officer, or scientific and technical police officer of the national police in France for more than a year, or work for the Ministry of the Interior as support staff, or medical staff,
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
To identify and describe the barriers and facilitators to the treatment of police officers facing mental health difficulties. | Up to 1 year
  * The analysis of the interviews with the police officers will be carried out using a method inspired by grounded theory; with first a deductive approach, then inductive; thirdly, links will be sought between the different categories of analysis to try to develop a synthetic representation of the barriers and facilitators to the treatment of police officers with mental health disorders.
  * Grounded theory research assumes that data, rather than existing theories or hypotheses, determine what knowledge is revealed. By systematically analyzing qualitative data, it seeks to understand the social phenomena studied.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pathologie Professionnelle - Médecine du Travail - CHU de Strasbourg - France, Strasbourg, France